CLINICAL TRIAL: NCT00678769
Title: Phase I Study of IMC-A12 (NSC# 742460) in Combination With Temsirolimus CCI-779 (NSC# 683864) in Patients With Advanced Cancers
Brief Title: Cixutumumab and Temsirolimus in Treating Patients With Locally Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00282; NCI-2009-00282 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000595388; 2007-0595 (Other: M D Anderson Cancer Center); 8109 (Other: CTEP); P30CA016672 (NIH); U01CA062461 (NIH); U01CA062487 (NIH); NCT00678223 (obsolete NCT alias)
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — cixutumumab; temsirolimus; Sirolimus

ARMS (3):
- Group A (temsirolimus on days 15 and 22 course 1) (Experimental): Patients receive temsirolimus IV over 30 minutes on days 15 and 22 for course 1 and on days 1, 8, 15, and 22 for all subsequent courses. Patients also receive cixutumumab IV over 60 minutes on days 1, 8, 15, and 22.
  Interventions: Drug: Cixutumumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Temsirolimus
- Group B (cixutumumab on days 15 and 22 of course 1) (Experimental): Patients receive cixutumumab IV over 60 minutes on days 15 and 22 for course 1 and on days 1, 8, 15, and 22 for all subsequent courses. Patients also receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
  Interventions: Drug: Cixutumumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Temsirolimus
- Group C (temsirolimus on days 1, 8, 15, and 22) (Experimental): Patients receive temsirolimus IV over 30 minutes and cixutumumab IV over 60 minutes on days 1, 8, 15, and 22.
  Interventions: Drug: Cixutumumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Temsirolimus

INTERVENTIONS:
Drug: Cixutumumab — Given IV
  Other Names: Anti-IGF-1R Recombinant Monoclonal Antibody IMC-A12; IMC-A12
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel

SUMMARY:
This phase I trial studies the side effects and best dose of cixutumumab and temsirolimus in treating patients with locally advanced or metastatic cancer. Monoclonal antibodies, such as cixutumumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Temsirolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving cixutumumab together with temsirolimus may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability; and to determine maximum tolerated dose (MTD) of the combination of IMC-A12 (cixutumumab) with temsirolimus in patients with or without biopsiable advanced cancers.

II. To evaluate the biologic effect of each individual drug and this drug combination on expression/phosphorylation of potential markers of response in patients with biopsiable disease.

III. To assess tumor metabolism by positron emission tomography (PET).

SECONDARY OBJECTIVES:

I. To report the clinical tumor response of this combination in a descriptive fashion.

OUTLINE:

DOSE ESCALATION PHASE: Patients receive temsirolimus intravenously (IV) over 30 minutes and cixutumumab IV over 60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. After the MTD is determined, subsequent patients are enrolled into the MTD expansion cohort.

MTD EXPANSION COHORT: Patients are assigned to 1 of 3 treatment groups.

GROUP A: Patients receive temsirolimus IV over 30 minutes on days 15 and 22 for course 1 and on days 1, 8, 15, and 22 for all subsequent courses. Patients also receive cixutumumab IV over 60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

GROUP B: Patients receive cixutumumab IV over 60 minutes on days 15 and 22 for course 1 and on days 1, 8, 15, and 22 for all subsequent courses. Patients also receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

GROUP C: Patients receive temsirolimus IV over 30 minutes and cixutumumab IV over 60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or metastatic cancer
* Patients enrolled in the expansion cohorts may be on antidiabetic treatment, but baseline glucose should be =< 120
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study; patients must also have signed an authorization for the release of their protected health information
* Patients are allowed to have unlimited prior treatments
* Patients must be registered in the MD Anderson Cancer Center (MDACC) institutional database (CORE) prior to treatment with study drug
* Estimated life expectancy of greater than 3 months
* Patients must be ≥ 4 weeks beyond treatment of any chemotherapy, other investigational therapy, biological, targeted agents or radiotherapy, and must have recovered to =< grade 1 toxicity or previous baseline for each toxicity; exceptions: patients must be >= 6 weeks beyond treatment with monoclonal antibodies; patients may have received palliative low dose radiotherapy to the limbs 1-4 weeks before this therapy provided pelvis, sternum, scapulae, vertebrae, or skull were not included in the radiotherapy field
* Patients must be >= 2 weeks beyond treatment of hormonal therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Absolute neutrophil count >= 1500/mL
* Platelets >= 100,000/mL
* Creatinine =< 2 X upper limit of normal (ULN)
* Total (T.) bilirubin =< 1.5 X ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and/or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5 X ULN
* Women of childbearing potential MUST have a negative serum or urine human chorionic gonadotropin (HCG) test unless prior hysterectomy or menopause (defined as 12 consecutive months without menstrual activity); patients should not become pregnant or breastfeed while on this study; sexually active patients must agree to use contraception prior to study entry, for the duration of study participation, and for 3 months after the last dose
* Patients must be >= 16 years of age; patients with Ewing's Sarcoma must be >= 14 years of age

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Patients who are pregnant or breastfeeding
* Patients with history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days
* Patients with uncontrolled intercurrent illness including, but not limited to, active infection requiring hospitalization
* Patients with history of hypersensitivity to monoclonal antibody treatment or immunosuppressant agents
* Patients with history of cerebrovascular accident (CVA), myocardial infarction or unstable angina within the previous six months before starting therapy
* Patients with New York Heart Association class III or greater congestive heart failure or uncontrolled hyperlipidemia (cholesterol > 300 mg/dl; triglyceride 2.5 X ULN despite lipid lowering agent)
* Patients with fasting blood sugar > 120; patients who are on oral hypoglycemic agents and insulin will be excluded; exception: patients in the expansion cohorts may be on antidiabetic treatment (including hypoglycemic agents and/or insulin) if controlled
* Patients on drugs that are strong P450 cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors or inducers; these drugs should be stopped 5 half-lives prior to starting investigational agents with temsirolimus; the strong inducing or inhibiting agents should not restart until 1 week after the end of study treatment; the principal investigator (PI) or his designee will go over/check the list of medication for individual patients; NOTE: Physiologic replacement of steroids (with either prednisone or hydrocortisone) in patients with adrenalectomy will be allowed
* Patients with history of brain metastasis are eligible, however the brain metastases should have been treated (treatment defined as surgery or radiation therapy [RT]) and the patient should have been free from symptoms/signs and off steroids for at least 3 months before study entry
* Patients with highly aggressive lymphoma (i.e. Burkitt's)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-05; Primary Completion 2013-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in phosphorylation levels of other biomarkers before and after treatment | Baseline to up to day 11
  Other markers include: insulin-like growth factor 1 receptor (IGF-1R), phosphorylated (p)IGF-1R, insulin receptor substrate-1 (IRS-1), phosphatase and tensin homolog gene (PTEN), vascular endothelial growth factor receptor (VEGFR)-1, VEGFR-2, and cluster of differentiation (CD)31. Generalized Estimating Equations model will be used to model the correlated IHC score between treatment arms.
Change in phosphorylation levels of v-akt murine thymoma viral oncogene homolog 1 in terms of difference in IHC score | Baseline to up to day 11
  Generalized Estimating Equations model will be used to model the correlated IHC score between treatment arms.
MTD of combination of cixutumumab and temsirolimus defined as the highest dose level at which no more than 1 of 6 evaluable patients has had a dose-limiting toxicity | 28 days
Tumor metabolism as assessed by PET scan before and after treatment | Baseline to up to day 28 of course 2
  The PET standardized uptake value (SUV) of all patients will be pooled together to plot the overall trend of PET SUV over time, the percent change in PET SUV will be estimated and 95% confidence intervals will be provided.

SECONDARY OUTCOMES:
Tumor response rate defined as CR + PR assessed by Response Evaluation Criteria in Solid Tumors and CHESON criteria | Up to 30 days after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Liu X, Lorusso P, Mita M, Piha-Paul S, Hong DS, Fu S, McQuinn L, Asatiani E, Doyle LA, Chen HX, Hess KR, Kurzrock R, Naing A. Incidence of mucositis in patients treated with temsirolimus-based regimens and correlation to treatment response. Oncologist. 2014 Apr;19(4):426-8. doi: 10.1634/theoncologist.2013-0231. Epub 2014 Mar 25. PMID 24668327